CLINICAL TRIAL: NCT03177070
Title: Investigating the Use of Fluorescent Imaging and Methylene Blue to Identify and Prevent Ureteric Injuries During Laparoscopic and Open Colorectal Surgery
Brief Title: Fluorescent Imaging & Methylene Blue: Ureter Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10871
Record Dates: First submitted 2017-05-15; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Ureteric Injury; Surgery; Surgery--Complications
Keywords: Ureteric injury; Colorectal Surgery
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methylene Blue (Experimental): Intravenous administration of methylene blue and assessment of ureteric fluorescence intraoperatively.
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue — As described above. Intravenous injection with visualisation via fluorescence enabled laparoscope.

SUMMARY:
The main aim of this project is to assess whether intravenous methylene blue can help identify the ureters during open and laparoscopic (keyhole) surgery. The ureters are small tubes that link the kidney to the bladder and, if not properly identified during surgery, may be damaged.

Methylene blue has been safely given to patients for many years and it is fluorescent. It is removed by the kidney and will therefore travel through the ureters. Methylene blue shines brightly (becomes fluorescent) when viewed under red light.

This study aims to compare the ability of methylene blue with white light to identify the location of the ureters during colorectal surgery. Recruitment will include 50 patients undergoing colorectal surgery (25 for keyhole/laparoscopic, 25 for open procedures). Each patient will act as their own control.

To detect the fluorescence, a special fluorescent laparoscope for keyhole surgery will be utilised, and a wide-field camera will be used for open surgery.

The potential benefits of this procedure are to identify the ureters during surgery and therefore prevent inadvertent damage to them

It is hoped that near infra-red light emitting from the ureters will be detected. This will allow the surgeon to determine the anatomy of the ureters during the operation and avoid inadvertent injury.

Funding source: Nuffield Department of Surgical Sciences, University of Oxford Recruitment sites: Oxford University Hospitals NHS Trust.

ELIGIBILITY:
Inclusion Criteria

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Patients undergoing laparoscopic or open colorectal surgery
* In the Investigator's opinion, is able and willing to comply with all study requirements.

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

* Patient who is unable or unwilling to give informed consent
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Significant renal or hepatic impairment.
* Any patients with previous allergies to Methylene Blue
* Any patients at risk of serotonin syndrome, including those taking serotonin reuptake inhibitors (SSRIs) or serotonin reuptake inhibitors (e.g. duloxetine, sibutramine, venlafaxine, clomipramine, imipramine)
* Patients with glucose-6-phosphate dehydrogenase (G6PD deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
To compare the change in ureter identification over time using white light versus intravenous methylene blue in each patient. | This will be assessed at the following time points post methylene blue administration: 0 minutes; 5 minutes; 10 minutes; 20 minutes; 30 minutes; 40 minutes; 50 minutes; 60 minutes; 70 minutes; 80 minutes; 90 minutes; 100 minutes.
  Ureter identification with and without fluorescence.

SECONDARY OUTCOMES:
Fluorescence quantification following administration of methylene blue between dosing cohorts post methylene blue administration. | This will be assessed at the following time points post methylene blue administration: 0 minutes; 5 minutes; 10 minutes; 20 minutes; 30 minutes; 40 minutes; 50 minutes; 60 minutes; 70 minutes; 80 minutes; 90 minutes; 100 minutes.
  Fluorescence quantification is measured using signal to background ratio. Signal is assessed on images using software that determines the brightness of a selected area using the average intensity of Red, Green and Blue pixels.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Yeung, MBChB, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD